CLINICAL TRIAL: NCT02559310
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Lefamulin (BC 3781) Versus Moxifloxacin (With or Without Adjunctive Linezolid) in Adults With Community-Acquired Bacterial Pneumonia
Brief Title: Study to Compare Lefamulin to Moxifloxacin (With or Without Linezolid) for the Treatment of Adults With Pneumonia
Acronym: LEAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAB-BC-3781-3101
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Community Acquired Pneumonia
Keywords: Pneumonia; CABP; CAP; Community acquired bacterial pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — lefamulin; Moxifloxacin; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lefamulin (Experimental): Intravenous lefamulin with potential step-down to oral lefamulin
  Interventions: Drug: lefamulin
- Moxifloxacin +/- Linezolid (Active Comparator): Intravenous moxifloxacin with potential step-down to oral moxifloxacin +/- linezolid
  Interventions: Drug: Moxifloxacin; Drug: Linezolid

INTERVENTIONS:
Drug: lefamulin — antibacterial agent
  Other Names: BC-3781
  Arms: Lefamulin
Drug: Moxifloxacin — antibacterial agent
  Other Names: Avelox
  Arms: Moxifloxacin +/- Linezolid
Drug: Linezolid — antibacterial agent
  Other Names: Zyvox
  Arms: Moxifloxacin +/- Linezolid

SUMMARY:
This study evaluates the safety and efficacy of lefamulin, a pleuromutilin, for the treatment of adults with moderate to severe community-acquired bacterial pneumonia.

DETAILED DESCRIPTION:
Lefamulin is a potent, semi-synthetic antibacterial belonging to a novel class known as the pleuromutilins. Both the intravenous (IV) and oral dosage forms of lefamulin are under investigation in this study. Lefamulin's in vitro antibacterial profile includes the most important bacterial pathogens causing respiratory tract infection (RTI). The antibacterial spectrum comprises S. pneumoniae, H. influenzae, M. catarrhalis, the atypical respiratory pathogens L. pneumophila, C. pneumoniae, and M. pneumoniae, S. aureus including MRSA and CA-MRSA, ß-haemolytic streptococci including S. pyogenes and S. agalactiae, and Enterococcus faecium including vancomycin-resistant enterococci (VRE). Moreover, as demonstrated in cross-resistance studies, lefamulin remains active against clinical isolates resistant to the following antimicrobial(s) (classes): macrolides, lincosamides, streptogramin B, oxazolidinones, tetracyclines, ß lactams, quinolones, trimethoprim-sulfametoxazole, mupirocin, and vancomycin.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female at least 18 years of age.
2. Provide written informed consent and be willing and able to adhere to the study-specified procedures and restrictions.
3. Have an acute illness (7 days duration) with at least 3 of the following symptoms consistent with a lower respiratory tract infection (new or worsening):

   * Dyspnea
   * New or increased cough
   * Purulent sputum production
   * Chest pain due to pneumonia
4. Have at least 2 of the following vital sign abnormalities:

   * Fever (body temperature >38.0°C (100.4°F) measured orally or equivalent temperature from an alternate body site) or hypothermia (body temperature <35.0°C (95.0°F) measured orally or equivalent temperature from an alternate body site)
   * Hypotension (systolic blood pressure <90 mmHg)
   * Tachycardia (heart rate >100 beats/min)
   * Tachypnea (respiratory rate >20 breaths/min)
5. Have at least 1 other clinical sign or laboratory finding of CABP:

   * Hypoxemia (i.e., O2 saturation <90% on room air or while receiving supplemental oxygen at subject's baseline requirement or PaO2 <60 mmHg)
   * Auscultatory and/or percussion findings consistent with pneumonia (e.g., crackles, egophony, dullness)
   * White blood cell (WBC) count >10,000 cells/mm3 or <4500 cells/mm3 or >15% immature neutrophils (bands) regardless of total WBC count
6. Have radiographically-documented pneumonia within 48 hours before enrollment (i.e., infiltrates in a lobar or multilobar distribution or diffuse opacities on chest x-ray or chest computed tomography scan consistent with acute bacterial pneumonia).
7. Have a Pneumonia Outcomes Research Team (PORT) Risk Class ≥III.

Exclusion Criteria:

1. Have received more than a single dose of a short-acting oral or IV antibacterial for CABP within 72 hours before randomization
2. Require concomitant systemic antibacterial therapy potentially effective against CABP pathogens
3. Have been hospitalized for 2 or more days within 90 days prior to the onset of symptoms or have resided in a nursing home or long-term healthcare facility within 30 days prior to the onset of symptoms. NOTE: Residence in an independent living facility is permitted.
4. Have confirmed or suspected CABP caused by a pathogen known to be resistant to any of the study drugs (e.g., Pseudomonas aeruginosa, any pathogen of the Enterobacteriaceae Family) or attributable to etiologies other than community acquired bacterial pathogens (e.g., ventilator associated pneumonia, hospital acquired bacterial pneumonia, bacterial aspiration pneumonia, Pneumocystis jiroveci pneumonia or other fungal pneumonia, viral or mycobacterial infection of the lung).
5. Have a noninfectious cause of pulmonary infiltrates (e.g., pulmonary embolism, chemical pneumonitis from aspiration, hypersensitivity pneumonia, congestive heart failure, bronchial obstruction, lung cancer, cystic fibrosis).
6. Have confirmed or suspected pleural empyema (does not include sterile parapneumonic effusions).
7. Require mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Schranz, MD, Study Chair — Nabriva Therapeutics
Locations (99):
- United States (7):
  - Site 1006, Hazard, Kentucky
  - Site 1008, Shreveport, Louisiana
  - Site 1005, Minneapolis, Minnesota
  - Site 1001, Butte, Montana
  - Site 1009, Akron, Ohio
  - Site 1002, Dayton, Ohio
  - Site 1004, Splendora, Texas
- Argentina (6):
  - Site 3005, La Plata, Buenos Aires
  - Site 3006, Rosario, Santa Fe Province
  - Site 3003, Córdoba
  - Site 3007, Córdoba
  - Site 3001, Córdoba
  - Site 3004, Córdoba
- Bosnia and Herzegovina (3):
  - Site 4003, Mostar
  - Site 4001, Tuzla
  - Site 4004, Zenica
- Brazil (4):
  - Site 3104, Belo Horizonte, Minas Gerais
  - Site 3102, Passo Fundo, Rio Grande Do Sol
  - Site 3103, Campinas, São Paulo
  - Site 3101, Sao Paulo Do Rio Preto, São Paulo
- Bulgaria (12):
  - Site 4105, Gabrovo
  - Site 4107, Lovech
  - Site 4112, Pernik
  - Site 4103, Rousse
  - Site 4108, Smolyan
  - Site 4102, Sofia
  - Site 4101, Sofia
  - Site 4106, Sofia
  - Site 4110, Sofia
  - Site 4111, Sofia
  - Site 4104, Veliko Tarnovo
  - Site 4109, Vidin
- Georgia (5):
  - Site 4206, Tbilisi
  - Site 4204, Tbilisi
  - Site 4205, Tbilisi
  - Site 4201, Tbilisi
  - Site 4202, Tbilisi
- Hungary (7):
  - Site 4305, Budapest
  - Site 4306, Csorna
  - Site 4304, Debrecen
  - Site 4302, Farkasgyepű
  - Site 4307, Miskolc
  - Site 4308, Miskolc
  - Site 4303, Törökbálint
- Latvia (3):
  - Site 4403, Daugavpils
  - Site 4401, Liepāja
  - Site 4402, Riga
- Netherlands (2):
  - Site 4603, Almelo, Overijssel
  - Site 4602, Helmond
- Peru (4):
  - Site 3205, Trujillo, La Libertad
  - Site 3202, Lima
  - Site 3204, Lima
  - Site 3201, Lima
- Philippines (5):
  - Site 2005, Iloilo City
  - Site 2003, Manila
  - Site 2004, Manila
  - Site 2002, Quezon City
  - Site 2001, Quezon City
- Poland (4):
  - Site 4703, Skierniewice, Lódzkie
  - Site 4704, Warsaw, Masovian Voivodeship
  - Site 4701, Lódz
  - Site 4702, Wilkowice
- Romania (9):
  - Site 4802, Palazu Mare, Constanța County
  - Site 4810, Bucharest
  - Site 4801, Bucharest
  - Site 4806, Bucharest
  - Site 4811, Cluj-Napoca
  - Site 4803, Craiova
  - Site 4808, Craiova
  - Site 4807, Timișoara
  - Site 4809, Timișoara
- Russia (6):
  - Site 4904, Chelyabinsk
  - Site 4902, Novosibirsk
  - Site 4903, Saint Petersburg
  - Site 4901, Saint Petersburg
  - Site 4906, Smolensk
  - Site 4905, Yaroslavl
- Serbia (4):
  - Site 5003, Niš, Nišavski Okrug
  - Site 5002, Belgrade
  - Site 5004, Kamenitz
  - Site 5001, Kragujevac, Šumadijski Okrug
- South Africa (5):
  - Site 5103, Benoni, Gauteng
  - Site 5104, Pretoria, Gauteng
  - Site 5105, Thabazimbi, Limpopo
  - Site 5101, Middelburg, Mpumalanga
  - Site 5102, Krugersdorp
- Site 2103, Nonthaburi, Thailand
- Ukraine (12):
  - Site 5203, Chernivtsi, Chernivtsi Oblast
  - Site 5204, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Site 5201, Kharkiv, Kharkivs’ka Oblast’
  - Site 5209, Kherson, Kherson Oblast
  - Site 5211, Odesa, Odesa Oblast
  - Site 5210, Zaporizhzhia, Zaporizhzhia Oblast
  - Site 5207, Kiyiv
  - Site 5202, Kyiv
  - Site 5205, Kyiv
  - Site 5208, Sumy
  - Site 5212, Zaporizhzhia
  - Site 5206, Zhytomyr

REFERENCES:
- [Derived] File TM Jr, Alexander E, Goldberg L, Das AF, Sandrock C, Paukner S, Moran GJ. Lefamulin efficacy and safety in a pooled phase 3 clinical trial population with community-acquired bacterial pneumonia and common clinical comorbidities. BMC Pulm Med. 2021 May 8;21(1):154. doi: 10.1186/s12890-021-01472-z. PMID 33964925
- [Derived] File TM, Goldberg L, Das A, Sweeney C, Saviski J, Gelone SP, Seltzer E, Paukner S, Wicha WW, Talbot GH, Gasink LB. Efficacy and Safety of Intravenous-to-oral Lefamulin, a Pleuromutilin Antibiotic, for the Treatment of Community-acquired Bacterial Pneumonia: The Phase III Lefamulin Evaluation Against Pneumonia (LEAP 1) Trial. Clin Infect Dis. 2019 Nov 13;69(11):1856-1867. doi: 10.1093/cid/ciz090. PMID 30722059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to enroll adults with CABP that was severe enough to require a minimum of at least 3 days of IV treatment. Subjects with a PORT score of III, IV and V were eligible. The first subject was randomized in February 2016 and the last subject was randomized in April 2017.
Pre-assignment Details: Subjects who met inclusion criteria and did not meet exclusion criteria were randomly assigned to a treatment group. Administration of study drug was expected to occur as soon as possible after the diagnosis of CABP with all Screening/Baseline assessments expected to be completed within 24 hours before the first dose IV study drug.
Groups:
- Lefamulin: Lefamulin 150 mg IV q12h with option to switch to 600 mg PO q12h after at least 6 doses of IV treatment. Linezolid placebo q12h was added at baseline for patients with suspected MRSA.
- Moxifloxacin ± Linezolid: Moxifloxacin 400 mg IV q24h with option to switch to 400 mg PO q24h after at least 6 doses of IV treatment. Linezolid 600 mg IV q12h was added at baseline for patients with suspected MRSA.
Period: Overall Study
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid
Started | 276 | 275
Completed | 249 | 256
Not Completed | 27 | 19
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Sponsor Decision | 0 | 1
Not completed — Randomized but not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid | Total
Number analyzed (Participants) | 276 | 275 | 551
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (16.31) | 59.6 (14.86) | 60.3 (15.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 160 | 330
  Male | 106 | 115 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 268 | 265 | 533
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 25 | 20 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 239 | 239 | 478
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 3 | 6 | 9
  Romania | 7 | 4 | 11
  Hungary | 10 | 13 | 23
  United States | 2 | 1 | 3
  Philippines | 23 | 17 | 40
  Ukraine | 55 | 61 | 116
  Thailand | 0 | 1 | 1
  Russia | 8 | 13 | 21
  Latvia | 17 | 11 | 28
  Netherlands | 1 | 0 | 1
  Brazil | 0 | 1 | 1
  Poland | 6 | 1 | 7
  South Africa | 12 | 15 | 27
  Georgia | 25 | 29 | 54
  Bulgaria | 65 | 58 | 123
  Serbia | 30 | 27 | 57
  Bosnia and Herzegovina | 11 | 14 | 25
  Peru | 1 | 3 | 4
Pneumonia Outcomes Research Team (PORT) Risk Class [Count of Participants; unit: Participants] — PORT Risk Class is a clinical prediction rule used to calculate risk of morbidity and mortality among patients presenting with community-acquired pneumonia taking into consideration age, history of comorbid conditions, physical examination findings, and laboratory or radiographic results. PORT Risk Class I is a PORT score of 0-50, II is 51-70, III is 71-90, IV is 91-130 and V is >130 with higher risk class indicating higher risk of morbidity and mortality.
  Participants
    II | 0 | 1 | 1
    III | 196 | 201 | 397
    IV | 76 | 70 | 146
    V | 4 | 3 | 7
CURB-65 Score [Count of Participants; unit: Participants] — CURB-65 is a clinical tool used to predict mortality in patients with community acquired pneumonia. The risk of death at 30 days increases as the score increases; a score of 0 indicates the lowest risk of death and a score of 5 indicates the highest risk of death. Defined as confusion of new onset, BUN >19 mg/dL, respiratory rate ≥30 breaths/min, systolic blood pressure <90 mm Hg or diastolic blood pressure ≤60 mm Hg, and age ≥65 years.
  Participants
    0 | 24 | 33 | 57
    1 | 130 | 121 | 251
    2 | 98 | 97 | 195
    3 | 22 | 22 | 44
    4 | 2 | 2 | 4
American Thoracic Society (ATS) Minor Severity Criteria [Count of Participants; unit: Participants] — ATS minor criteria are used to indicate severe community acquired pneumonia and suggests the need for intensive care unit (ICU) level care. Defined as presence of 3 or more of the following 9 criteria at baseline: respiratory rate of 30 breaths/min or greater, oxygen saturation less than 90% or PaO2 less than 60mmHg, blood urea nitrogen level of 20mg/dL or greater, white blood cell count less than 4,000/mm3, confusion, multilobar infiltrates, platelet level less than 100,000 cells/mm3, temperature lower than 36 °C, or systolic blood pressure less than 90mmHg.
  Participants | 54 | 48 | 102
Systemic inflammatory response syndrome (SIRS) Criteria [Count of Participants; unit: Participants] — SIRS is used to define a clinical response to a nonspecific insult of either infectious or noninfectious origin. SIRS is defined as a subject meeting at least 2 or more of the following: Fever of more than 38C (100.4F) or less than 36C (96.8F); heart rate greater than 90 beats/min; respiratory rate greater than 20 breaths/min or PaCO2 less than 32 mm Hg; abnormal white blood cell count (greater than 12,000/microL or less than 4,000/microL or greater than 10% immature band forms)
  Participants | 268 | 267 | 535
Bacteremic [Count of Participants; unit: Participants] | 7 | 3 | 10
Received Single Dose Short Acting Systemic Antibacterial within 72 hrs of Randomization [Count of Participants; unit: Participants] | 66 | 66 | 132
Renal Status [Count of Participants; unit: Participants]
  Severe Impairment (CrCl <30mL/min) | 3 | 3 | 6
  Moderate Impairment (CrCl 30-<60mL/min) | 61 | 62 | 123
  Mild Impairment (CrCl 60-<90mL/min) | 89 | 75 | 164
  Normal Function (CrCl >=90mL/min) | 121 | 134 | 255
  Missing renal status | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response (ECR)
Description: ECR was defined as survival with improvement in at least 2 signs and symptoms of CABP (relative to baseline), no worsening of any CABP sign or symptom, and no use of concomitant antibiotics (other than adjunctive linezolid, as allowed by the study protocol) for the treatment of CABP through the ECR assessment.
Time Frame: ECR was assessed 96 +/- 24 hours after the first dose of study drug.
Population: Intent to Treat Analysis Set: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid
Number analyzed (Participants) | 276 | 275
Participants
  Responder | 241 | 248
  Non-Responder | 29 | 21
  Indeterminate | 6 | 6
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin ± Linezolid; Test type: Non-Inferiority — Non-inferiority Margin = 12.5%; Treatment Difference (Lef - Mox) = -2.9, 95% CI 2-sided [-8.5 to 2.8] — Difference in percentage of Responders for ECR (Lefamulin - Moxifloxacin). CI computed using continuity-corrected Z-statistic

2. Secondary Outcome: Investigator's Assessment of Clinical Response (IACR)
Description: IACR was defined as resolution or improvement of a subject's clinical signs and symptoms such that no additional antibacterial therapy was administered for the treatment of the current episode of CABP
Time Frame: IACR was assessed at the Test-of-Cure visit; 5-10 days after the last dose of study drug.
Population: Modified ITT population: All randomized subjects who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid
Number analyzed (Participants) | 273 | 273
Participants
  Success | 223 | 230
  Failure | 43 | 40
  Indeterminate | 7 | 3
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin ± Linezolid; Test type: Non-Inferiority — Non-inferiority Margin = 10%; Treatment Difference (Lef - Mox) = -2.6, 95% CI 2-sided [-8.9 to 3.9] — Difference in Percentage of Success for IACR at test of cure visit (Lefamulin - Moxifloxacin). CI computed via Miettinen-Nurminen method, adjusted for prior antibiotic use [Y vs. N] and PORT risk class [III vs. IV/V], using CMH stratum weights
Statistical Analysis 2: Comparison: Lefamulin; Test type: Non-Inferiority — Non-Inferiority Margin = 10%; Treatment Difference (Lef - Mox) = -2.6, 95% CI 2-sided [-9.2 to 4.1] — Difference in percentage of Success for IACR at test of cure visit. CI computed using continuity-corrected Z-statistic

3. Secondary Outcome: Investigator's Assessment of Clinical Response (IACR)
Description: as for outcome 2
Time Frame: IACR was assessed at the Test of Cure visit, 5 - 10 days after the last dose of study drug.
Population: Clinically Evaluable population: Subset of ITT population having met additional pre-defined criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid
Number analyzed (Participants) | 236 | 245
Participants
  Success | 205 | 219
  Failure | 31 | 26
Statistical Analysis 1: Comparison: Lefamulin vs Moxifloxacin ± Linezolid; Test type: Non-Inferiority — Non-Inferiority Margin = 10%; Treatment Difference = -2.5, 95% CI 2-sided [-8.4 to 3.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Lefamulin vs Moxifloxacin ± Linezolid; Test type: Non-Inferiority — Non-Inferiority Margin = 10%; Treatment Difference (Lef - Mox) = -2.5, 95% CI 2-sided [-8.7 to 3.7] — Difference in Percentage of Success for IACR at test of cure visit (Lefamulin - Moxifloxacin). CI computed using continuity-corrected Z-statistic

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of informed consent through the completion of the Test-of-Cure (TOC) Visit (i.e., 5-10 days after the last dose of study drug). Serious adverse events were recorded from the time of informed consent to the Late Follow-Up Visit (approximately 30 days after the first dose of study drug).
Description: Adverse events are reported for randomized subjects who received at least one dose of study drug (Safety Population). Treatment-emergent adverse events, defined as events occurring after the first dose of study drug, are reported. Adverse events were recorded whether or not they were considered to be study drug related.
Arm/Group | Lefamulin | Moxifloxacin ± Linezolid
All-Cause Mortality (participants affected / at risk) | 6/273 | 5/273
Serious Adverse Events (participants affected / at risk) | 19/273 | 13/273
Other Adverse Events (participants affected / at risk) | 39/273 | 46/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lefamulin (N=273) | Moxifloxacin ± Linezolid (N=273)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Injection Site Reaction (General disorders) | 1 | 0
Infectious Pleural Effusion (Infections and infestations) | 1 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Viral Pharyngitis (Infections and infestations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular Seminoma (Pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lefamulin (N=273) | Moxifloxacin ± Linezolid (N=273)
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 8 | 6
Insomnia (Psychiatric disorders) | 8 | 5
Infusion Site Pain (General disorders) | 8 | 0
Infusion Site Phlebitis (General disorders) | 6 | 3
Alanine Aminotransferase Increased (Investigations) | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 21
Hypertension (Vascular disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data from the study is confidential information. Sponsor has the right to publish first. Thereafter, PI may publish data from the study, but PI must submit the publication to Sponsor for review at least 60 days prior to publication. Sponsor may remove any confidential and/or proprietary information. If Sponsor's publication is not submitted within 12 months after the study, or if Sponsor decides not to publish, PI may publish the data, subject to Sponsor's rights in the agreement.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02559310/SAP_000.pdf
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02559310/Prot_001.pdf